CLINICAL TRIAL: NCT05426681
Title: Spinal Cord Injury Neuroprotection With Glyburide (SCING): Pilot Study: An Open-Label Prospective Evaluation of the Feasibility, Safety, Pharmacokinetics, and Preliminary Efficacy of Oral Glyburide (DiaBeta) in Patients With Acute Traumatic Spinal Cord Injury
Brief Title: Spinal Cord Injury Neuroprotection With Glyburide
Acronym: SCING
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, Francis Farhadi, Associate Professor of Neurosurgery, University of Kentucky
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 77662
Record Dates: First submitted 2022-06-13; First posted 2022-06-22 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Acute Spinal Cord Injury
MeSH Terms: interventions — Glyburide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Glyburide treatment arm (Experimental)
  Interventions: Drug: GlyBURIDE Oral Tablet

INTERVENTIONS:
Drug: GlyBURIDE Oral Tablet — Enrolled patients will receive 12 doses of Glyburide starting within 8 hours of spinal cord injury. The dosing regimen involves an initial dose of 1.25mg followed by 11 consecutive doses of 0.625 mg every 6 hours. The total daily dose of Glyburide on Day 1, Day 2, and Day 3 will be 3.125 mg, 2.5 mg, and 2.5 mg respectively.
  Intervention: Drug: Glyburide
  Other Names: Diabeta

SUMMARY:
To assess the safety and efficacy of using oral Glyburide (Diabeta) as a neuroprotective agent in patients with acute cervical or thoracic traumatic spinal cord injury.

DETAILED DESCRIPTION:
This study will include subjects between 18 and 80 years who have experienced acute traumatic cervical or thoracic spinal cord injury. Subjects will begin an oral drug regimen of Glyburide with the initial dose being within 8 hours of the injury and again every 6 hours after for 72 total hours of treatment. The daily dose of 3.125mg on day one and 2.5 mg on days 2 and 3 will be used to determine if the investigational drug provides any neuroprotection when given soon after injury. If indicated, the subject will also have surgical intervention for spinal cord decompression surgery and spinal stabilization. Participants will have labs drawn regularly, and ECGs done throughout their hospital stay. Adverse events will be monitored daily through day 14 of participation or hospital discharge (whichever is earlier). Study participation will last for 365 days (+/- 30 days), with post-hospitalization follow-up occurring on days 28, 42, 84, 182, and 365.

ELIGIBILITY:
Inclusion Criteria:

* No life threatening injuries resulting from the traumatic accident
* No evidence of sepsis
* Acute cervical or thoracic SCI with ASIA Impairment Scale Grade A, B, or C od admission.
* Non-penetrating SCI at neurologic level from C2 to C8 or T1 to T12

Exclusion Criteria:

* Unconsciousness or other mental impairment that prevents neurological assessment within the first 8 hours
* Acute SCI with ASIA Impairment Scale grade D or E
* Currently involved in another non-observational SCI research study or receiving another investigational drug
* History of hypersensitivity to sulfonylureas, in particular glyburide, or any of its components
* Any condition likely to result in the patient's death within the next 12 months
* Severe renal disorder from the patient's history (e.g. dialysis) or baseline eGFR of < 30 mL/min/1.73 m2
* Known severe liver disease, or ALT > 3 times upper limit of normal or bilirubin
* Blood glucose <55 mg/dL at enrollment or immediately prior to administration of DiaBeta, or a clinically significant history of hypoglycemia
* Acute ST elevation myocardial infarction, and/or acute decompensated heart failure, and/or QTc > 520 ms, and/or known history of cardiac arrest (PEA, VT, VF, asystole), and/or admission for an acute coronary syndrome, myocardial infarction, or coronary intervention (percutaneous coronary intervention or coronary artery surgery) within the past 3 months
* Known G6PD enzyme deficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Rate of recruitment of patients with tSCI within the specified time window. | within 8 hours of tSCI
  A measure of feasibility of undertaking a large phase II study among this population of patients where treatment must begin within a short injury-to-drug time window.
Number of drug related adverse events. | One year post treatment
  A measure of safety of treating patients with traumatic spinal cord injury with Glyburide administered orally.

SECONDARY OUTCOMES:
Neurologic recovery following tSCI | One year post enrollment.
  Neurologic status be assessed using the American Spinal Injury Association Impairment Scale. This neurological exam assesses sensory and motor impairments using touch and pin prick evaluations in each dermatome and muscle strength. Right and left body sides are evaluated independently. Lower the scores indicate greater degree of impairment.
  Touch and pin prick perception is scored using a 0-2 and NT grade. Where 0= Absent, 1= hypo/hypersensitivity, 2= normal sensation, and NT= not testable. Scores for each body side are added together and summed for a total sensation score. Maximum score possible for this section is 112 per side.
  Muscle function is rated on a 0-5 scale. Where 0= total paralysis, 1= palpable/visible contraction, 2= active movement, full ROM with gravity eliminated, 3= active movement, full ROM against gravity, 4= active movement, full ROM with moderate resistance, 5= Normal movement and strength, and NT= not tested. Maximum score for this section is 50 per side.
Serum Pharmacokinetics to measure Glyburide concentrations. | Enrollment through post-treatment day 7.
  Plasma concentrations of Glyburide will be serially quantified through day 3 following tSCI to evaluate the pharmacokinetics of the investigational drug. Comparisons will be made to reported levels achieved in healthy patient cohorts.
Biomarker Analysis | Enrollment, Day 3, and Day 7
  Standard enzyme-linked immunosorbent assay (ELISA) techniques will be used to measure blood levels of neurofilament light chain, neuron- specific enolase, tau, S100b, and glial fibrillary acidic protein levels on admission, at 24 hours and on days 3 and 7 following tSCI to evaluate serum biomarker levels. Comparisons will be made to previously published values observed in non-treated control patients

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided